CLINICAL TRIAL: NCT02093481
Title: Intrinsic Indigestible Carbohydrates as Means to Modulate Colonic Events, With Specific Focus on Metabolism and Satiety
Brief Title: Effects of Dietary Fibre on Glucose Metabolism and Satiety
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Jonna Sandberg, MSc, postgraduate student, Lund University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Dnr2013/241
Record Dates: First submitted 2014-03-10; First posted 2014-03-21 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Obesity; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- + ind. CHO + prim (Experimental): Test meal: ate intrinsic indigestible carbohydrates 3 days prior to measurements of variables (priming)
  Interventions: Other: Test meal; Other: Priming
- - ind. CHO + prim (Experimental): Reference:ate no intrinsic indigestible carbohydrates 3 days prior to measurements of variables (priming)
  Interventions: Other: Reference; Other: Priming
- + ind. CHO - prim (Experimental): Test meal: ate intrinsic indigestible carbohydrates 1 day prior to measurements of variables (no priming)
  Interventions: Other: Test meal; Other: No priming
- - ind. CHO - prim (Experimental): Reference: ate no indigestible carbohydrates the day prior to measurements of variables (no priming).
  Interventions: Other: Reference; Other: No priming

INTERVENTIONS:
Other: Test meal
  Arms: + ind. CHO + prim; + ind. CHO - prim
Other: Reference
  Arms: - ind. CHO + prim; - ind. CHO - prim
Other: Priming — The reference or test meal was eaten 3 days prior to measurements of variables.
  Arms: + ind. CHO + prim; - ind. CHO + prim
Other: No priming — The reference or test meal was eaten 1 days prior to measurements of variables.
  Arms: + ind. CHO - prim; - ind. CHO - prim

SUMMARY:
The experimental model is a semi-acute study where the purpose of the study is to evaluate food factors related to colonially derived regulation of glucose metabolism (and related parameters) and satiety in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Normal fasting blood glucose, BMI 19-25 kg/m2

Exclusion Criteria:

* Gastrointestinal diseases or food allergies e.g. lactose-, gluten intolerance, metabolic disorders e.g. diabetes, tobacco/snuff users. Antibiotic or probiotic usage within two weeks, and during study. Vegetarians.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Blood glucose | Postprandial 0-180 min after breakfast
  The test products are both ingested one day and three days prior to measurements of variables.
Insulin | Postprandial 0-180 min after breakfast
  The test products are both ingested one day and three days prior to measurements of variables.
Appetite hormones | Postprandial 0-180 min after breakfast
  The test products are both ingested one day and three days prior to measurements of variables.
Markers of colonic fermentation and inflammation | Postprandial 0-180 min after breakfast
  The test products are both ingested one day and three days prior to measurements of variables.

SECONDARY OUTCOMES:
Subjective satiety | Postprandial 0-180 min after breakfast
  The measures of hunger, satiety, and desire to eat with the use of a VAS were determined every hour throughout the postprandial testing sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Nilsson, PhD, Principal Investigator — Lund Univeristy
Locations (1):
- Applied Nutrition and Food Chemistry, Lund Univeristy, Lund, SE, Sweden

REFERENCES:
- [Derived] Sandberg JC, Bjorck IM, Nilsson AC. Rye-Based Evening Meals Favorably Affected Glucose Regulation and Appetite Variables at the Following Breakfast; A Randomized Controlled Study in Healthy Subjects. PLoS One. 2016 Mar 18;11(3):e0151985. doi: 10.1371/journal.pone.0151985. eCollection 2016. PMID 26990559